CLINICAL TRIAL: NCT06396403
Title: The Role of Red Cell Characteristics, Angiogenesis, Viscosity and Oxygenation in the Pathophysiology of Sickle Cell Related Retinopathy
Acronym: RAVOS
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Bart J. Biemond, Prof. Dr. B.J. Biemond, MD PhD, Amsterdam UMC, location AMC
Other Study IDs: NL81111.018.22
Record Dates: First submitted 2024-04-24; First posted 2024-05-02 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Sickle Cell Retinopathy; Sickle Cell Disease; Sickle Cell SC Disease; Sickle Cell-SS Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — venous blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- HbSS patients without SCR: Adult sickle cell patients with the HbSS genotype and without sickle cell retinopathy
  Interventions: Other: Collection of venous blood samples
- HbSS patients with PSCR: Adult sickle cell patients with the HbSS genotype and proliferative sickle cell retinopathy
  Interventions: Other: Collection of venous blood samples
- HbSC patients without SCR: Adult sickle cell patients with the HbSC genotype and without sickle cell retinopathy
  Interventions: Other: Collection of venous blood samples
- HbSC patients with PSCR: Adult sickle cell patients with the HbSC genotype and proliferative sickle cell retinopathy
  Interventions: Other: Collection of venous blood samples

INTERVENTIONS:
Other: Collection of venous blood samples — collection includes 1 EDTA tube and 1 Sarstedt S-Monovette tube of 5 mL

SUMMARY:
Objective:

to gain insight in the pathogenesis, to identify biomarkers to recognize patients at risk for proliferative SCR and to investigate its associations with clinical and laboratory characteristics.

Endpoints:

The investigators will determine the difference in the above named parameters between patients with and without PSCR

Study design:

This case control study will include adult sickle cell disease patients with the HbSS or HbSC genotype. For both genotypes, 20 patients without sickle cell retinopathy (SCR) and 20 patients with PSCR will be included, resulting in a total of 80 patients. Venous blood samples and retinal imaging scans will be collected for each included patient.

DETAILED DESCRIPTION:
Rationale:

Sickle cell disease (SCD) is characterized by chronic hemolysis and recurrent microvascular occlusion, resulting in ischemia and organ damage1. This study focuses on retinal damage: sickle cell retinopathy (SCR). SCR results from ischemic vascular disease and secondary angiogenesis, but it is unknown which factors play a significant role in the pathogenesis. Studies on this subject are still in an early phase3,4. Our aim is to gain insight in the pathogenesis, to identify biomarkers to recognize patients at risk for proliferative SCR and to investigate its associations with clinical and laboratory characteristics. The focus of our study is aimed at evaluation of innovative biomarkers of angiogenesis, whole blood viscosity and innovative characterization of red blood cell parameters such as deformability, adhesiveness and "point of sickling" as can be measured ex vivo by the Oxygenscan (i.e.: red cell sickling capacity). The Oxygenscan is a new method to calculate the deformability of red blood cells as a function of the partial pressure of oxygen. These novel parameters will be related to clinical characteristics observed in these patients and specific markers of early retinopathy such as vessel density and macula thinning assessed by OCT angiography.

Objective:

The objective of this study is to gain insight in the pathogenesis, to identify the role of red cell characteristics, markers of angiogenesis, retinal oxygenation and whole blood viscosity in the development of proliferative SCR and to investigate its associations with clinical and laboratory characteristics.

Study design:

Case control study

Study population:

Adult patients with sickle cell disease (SCD) with a HbSS or HbSC genotype. For both genotypes, 20 patients without SCR and 20 patients with proliferative SCR will be included. The total amount of included patients will be 80 patients.

Intervention:

venous blood samples (1 EDTA tube and 1 PECT tubes of 4-5 mL each) will be collected from all included patients, who will be requested to fast 8 hours before the collection of blood. If fasting is not desired/possible, a low-fat breakfast can be consumed.

Main study parameters/endpoints: (1) The difference in red blood cell characteristics (point of sickling) between patients with and without PSCR, (2) The difference in plasma levels of parameters representing the level of systemic angiogenesis activity (CD105, VEGF, CTGF and angiopoietin-2) between patients with and without PSCR, (3) The difference in oxygenation of the retina by assessing the vessel density with angio-OCT and by assessing the oxygen saturation in the retinal arterioles and venules with the Oxymap scan in patients with and without PSCR, (4) The difference in whole blood viscosity between patients with and without PSCR

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Data from recent ophthalmologic and hematologic examinations will be collected. If no recent ophthalmologic examination is available and no further appointments were made yet, the patient will be contacted to visit the outpatient clinic for a new appointment. Since the appointments are in accordance with the general screening schedule according to the Dutch Guidelines for Sickle Cell Disease, these investigations are no extra burden for the patients. Venous blood samples will be obtained by venepuncture, preferably during the routine venepuncture for scheduled hematological visits (so the only extra burden consists of the extra blood aliquots that have be drawn to answer the research questions). Venepuncture is a safe and frequently used procedure in the routine care of patients with sickle cell disease. Due to the request to fast before the venepuncture, appointments will only be scheduled in the morning in order to reduce the burden on the patient as much as possible.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years
* HbSC or HbSS genotype
* Recent ophthalmologic examination (up to 2 years prior) or (willingness to attend) upcoming examination

Exclusion Criteria:

* Age below 18 years
* Genotype other than HbSC or HbSS
* No recent ophthalmologic examination and no intention to visit the outpatient clinic for ophthalmic and hematologic examination
* Participation in trials with either crizanlizumab, voxelotor or mitapivat.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with sickle cell disease (SCD) with the HbSS or HbSC genotype, attending the outpatient Sickle Cell Clinic from the Amsterdam UMC.
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2023-06-13 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-06-17 (Actual)

PRIMARY OUTCOMES:
Differences in Red blood cell characteristics (Oxygenscan) | Immediately after the venepuncture
  The difference in red blood cell characteristics (point of sickling) between patients with and without PSCR in both genotypes
Differences in Angiogenesis biomarkers | Immediately after the venepuncture
  The difference in plasma levels of parameters representing the level of systemic angiogenesis activity (CD105, VEGF, CTGF and angiopoietin-2) between patients with and without PSCR in both genotypes
Differences in Retinal Oxygenation | Immediately after the venepuncture
  The difference in oxygenation of the retina by assessing the vessel density with angio- OCT and by assessing the oxygen saturation in the retinal arterioles and venules with the Oxymap scan in patients with and without PSCR in both genotypes
Differences in Whole blood viscosity | Immediately after the venepuncture
  The difference in whole blood viscosity between patients with and without PSCR in both genotypes

SECONDARY OUTCOMES:
Associations between Oxygenation parameters and Red blood cell characteristics | Immediately after the venepuncture
  Association between retinal vessel density assessed by OCT-angiography, oxygen saturation assessed by an Oxymap scan and red blood cell characteristics (deformity, adhesion and point of sickling upon hypoxia)
Associations between sex, age, and genotype and the biomarkers of angiogenesis | Immediately after the venepuncture
  Association between sex, age, and genotype and the biomarkers of angiogenesis
Association between hemoglobin, and HbF and biomarkers of angiogenesis | Immediately after the venepuncture
  Association between hemoglobin, and HbF and biomarkers of angiogenesis
Associations between whole blood viscosity and genotype | Immediately after the venepuncture
  Associations between whole blood viscosity and genotype

CONTACTS AND LOCATIONS:
Overall Officials: Bart J Biemond, MD PhD, Principal Investigator — Department of Hematology, Amsterdam UMC, Amsterdam, The Netherlands
Locations (1):
- Amsterdam UMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No